CLINICAL TRIAL: NCT03674281
Title: The VRIF Trial: Hypoglycemia Reduction With Automated-Insulin Delivery System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Virginia (Other)
Collaborators: Virginia Research Investment Fund (Other); DexCom, Inc. (Industry); Tandem Diabetes Care, Inc. (Industry)
Responsible Party: Principal Investigator, Sue Brown, Associate Professor, University of Virginia
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 20964; VRIF-FY18-002 (Other Grant/Funding Number: Virginia Research Investment Fund)
Record Dates: First submitted 2018-09-14; First posted 2018-09-17 (Actual); Results first posted 2021-01-12 (Actual); Last update posted 2021-01-12 (Actual); Status verified 2020-12

CONDITIONS: Type 1 Diabetes Mellitus; Cognitive Change
Keywords: Closed-Loop Control (CLC); Sensor-Augmented Therapy (SAP); Insulin Pump; Artificial Pancreas (AP); Continuous Glucose Monitor (CGM)
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Sensor Augmented Pump (SAP)-Closed-Loop Control (CLC) (Experimental): SAP: Subjects will be utilizing their own insulin pumps (without automated insulin delivery) plus Dexcom G6 CGM to control their blood glucose for 4 weeks. Subjects will be evaluated by actigraphy watch and by Ecological Momentary Assessments in approximately the final 14 days of the 4 week period.
  CLC with Control-IQ plus CGM: Following SAP, subjects will be utilizing the Tandem t:slim X2 with Control-IQ along with a Dexcom G6 continuous glucose monitor to control their blood glucose for 4 weeks. Subjects will be evaluated by actigraphy watch and by Ecological Momentary Assessments in approximately the final 14 days of the 4 week period.
  Interventions: Device: SAP; Device: CLC

INTERVENTIONS:
Device: SAP — Subjects will wear their own personal insulin pump and will wear the study CGM (Dexcom G6).
  Other Names: Sensor-augmented Pump
Device: CLC — The Tandem t:slim X2 is an insulin pump with software (Control-IQ Technology) that helps regulate blood glucose more optimally, based on data received from the Dexcom G6 CGM.
  Other Names: Tandem t:slim X2 with Control-IQ and Dexcom G6 CGM

SUMMARY:
The objective of this pilot study is (i) to test the use of an Artificial Pancreas (AP) System as a viable therapy treatment for two vulnerable populations: 6 to 10 year-old and adults older ≥65 years old with T1D; (ii) to assess cognitive function in children and older adult patients with T1D and examine whether improved glycemic control defined by stable (more than 70% of the day in glycemic range 70-180 mg/dL) control positively influences cognitive function; and (iii) obtain preliminary data to apply to funds to continue with larger and longer clinical trials.

DETAILED DESCRIPTION:
This study will evaluate up to 15 subjects in each age group for a period of 8-10 weeks performing neurocognitive tests before and after each intervention. The first study phase will be up to 2 weeks of a training period to allow participants to get acquainted with the use of the CGM if they are not familiar with the use of the device. This training period will be followed by a 4-week sensor-augmented pump (SAP) period using a study CGM and the subject's personal insulin pump. The subjects will return to clinic at the completion of the SAP period and will be trained on the Tandem t:slim X2 with Control-IQ and G6 CGM. At the completion of the system training session, subjects will begin 4-weeks of Closed-Loop Control (CLC). Questionnaires will be completed by the study subject at screening, after completion of SAP and after completion of CLC. Ecological Momentary Assessments (EMAs) and actigraphy data will be collected in the last 14 days of the SAP and CLC periods.

A parent/guardian of the enrolled children will also be asked to participate in all trainings, complete parental Patient-Report Outcomes (PRO) Questionnaires, and collect sleep patterns while wearing the actigraph watch.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis, based on investigator assessment, of type 1 diabetes for at least one year, using insulin for at least 1 year and using an insulin pump for at least 6 months.
* Familiarity and use of a carbohydrate ratio for meal boluses by participants and families participating.
* Age 6-10 years old or 65 years or older
* Hemoglobin A1c <10%
* For females of child-bearing potential, not currently known to be pregnant:

A negative serum or urine pregnancy test will be required for all females of child-bearing potential. Participants who become pregnant will be discontinued from the study. Also, participants who during the study develop and express the intention to become pregnant within the timespan of the study will be discontinued.

* For participants <18 years old, living with one or more parent/legal guardian knowledgeable about emergency procedures for severe hypoglycemia and able to contact the participant in case of an emergency.
* Willing to disable any automated insulin delivery functionality on a personal insulin pump during study, such as Medtronic 670G in auto mode. Predictive low blood glucose suspend, such as Tandem insulin pump with Basal-IQ, will be allowed.
* Investigator has confidence that the participant and family can successfully operate all study devices and is capable of adhering to the protocol.
* Willingness to switch to lispro (Humalog) or aspart (Novolog) and to use no other insulin besides lispro (Humalog) or aspart (Novolog) during the study.
* Total daily insulin dose (TDD) at least 10 U/day.
* Willingness not to start any new non-insulin glucose-lowering agent during the course of the trial

Exclusion Criteria:

* Severe hypoglycemia resulting in seizure or loss of consciousness in the 12 months prior to enrollment.
* Diagnosis of Diabetic Ketoacidosis in the 12 months prior to enrollment.
* Uncontrolled cardiac disease (e.g. recent myocardial infarction, severe congestive heart failure).
* Cerebrovascular accident in the 12 months prior to enrollment.
* Uncontrolled resting arterial hypertension (>160/90 mm Hg).
* Conditions that would make use of a CGM difficult (e.g., blindness, severe arthritis, immobility).
* Current use of oral/inhaled glucocorticoids or other medications, which in the judgment of the investigator would be a contraindication to participation in the study.
* Concurrent use of any non-insulin glucose-lowering agent other than metformin (including GLP-1 agonists, pramlintide, DPP-4 inhibitors, SGLT-2 inhibitors, sulfonylureas).
* Hemophilia or any other bleeding disorder
* A condition, which in the opinion of the investigator or designee, would put the participant or study at risk
* Participation in another pharmaceutical or device trial at the time of enrollment or during the study
* Employed by, or having immediate family members employed by Tandem Diabetes Care, Inc., or having a direct supervisor at place of employment who is also directly involved in conducting the clinical trial (as a study investigator, coordinator, etc.); or having a first-degree relative who is directly involved in conducting the clinical trial.

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2018-09-24 (Actual); Primary Completion 2019-11-21 (Actual); Study Completion 2019-11-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sue Brown, MD, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: Yes
Will follow the NIH Data Sharing Policy and Implementation Guidance on sharing research resources for research purposes to qualified individuals within the scientific community.
Supporting Information: Study Protocol, ICF
Time Frame: Generally after publications are complete.
Access Criteria: Will follow data sharing policy.

RESULTS

PARTICIPANT FLOW:
Groups:
- Older Adults:Sensor Augmented Pump (SAP)-Closed-Loop Control (CLC); Younger Children: SAP-CLC: SAP: Subjects will be utilizing their own insulin pumps (without automated insulin delivery) plus Dexcom G6 CGM to control their blood glucose for 4 weeks. Subjects will be evaluated by actigraphy watch and by Ecological Momentary Assessments in approximately the final 14 days of the 4 week period.
  CLC with Control-IQ plus CGM: Following SAP, subjects will be utilizing the Tandem t:slim X2 with Control-IQ along with a Dexcom G6 continuous glucose monitor to control their blood glucose for 4 weeks. Subjects will be evaluated by actigraphy watch and by Ecological Momentary Assessments in approximately the final 14 days of the 4 week period.
  SAP: Subjects will wear their own personal insulin pump and will wear the study CGM (Dexcom G6).
  CLC: The Tandem t:slim X2 is an insulin pump with software (Control-IQ Technology) that helps regulate blood glucose more optimally, based on data received from the Dexcom G6 CGM.
- Parents of Young Children: Parent of Young Children. Parents wore a sleep watch.
Period: Overall Study
Arm/Group | Older Adults:Sensor Augmented Pump (SAP)-Closed-Loop Control (CLC) | Younger Children: SAP-CLC | Parents of Young Children
Started | 18 | 16 | 16
Completed | 15 | 13 | 13
Not Completed | 3 | 3 | 3
Not completed — screen failure | 2 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- Parents of Young Children: Limited data were obtained on parents of young children and included actigraphy watch.
- Total: Total of all reporting groups
Arm/Group | Older Adults:Sensor Augmented Pump (SAP)-Closed-Loop Control (CLC) | Younger Children: SAP-CLC | Parents of Young Children | Total
Number analyzed (Participants) | 15 | 13 | 13 | 41
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.7 (3.3) | 9.1 (0.9) | 42.9 (4.5) | 41.6 (25.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 8 | 12 | 26
  Male | 9 | 5 | 1 | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 1
  White | 14 | 13 | 13 | 40
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 15 | 13 | 13 | 41
Hemoglobin A1c [Mean (Standard Deviation); unit: percentage of glycosylated hemoglobin] | 7 (0.8) | 7.6 (1.2) | NA (NA) — Not obtained as it was not an enrollment criterion these participants. | 7.3 (1.0)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Time of Blood Glucose in Range 70-180 mg/dL
Description: Percentage of time of blood glucose in range 70-180 mg/dL as measured by the continuous glucose monitor.
Time Frame: One month during each study period (sensor augmented pump and closed loop control)
Measure: Mean (Standard Deviation); unit: percentage of time
Groups:
- Older Adults:Sensor Augmented Pump (SAP); Young Children: SAP: SAP: Subjects will be utilizing their own insulin pumps (without automated insulin delivery) plus Dexcom G6 CGM to control their blood glucose for 4 weeks. Subjects will be evaluated by actigraphy watch and by Ecological Momentary Assessments in approximately the final 14 days of the 4 week period.
- Older Adults: Closed-Loop Control (CLC); Young Children: CLC: CLC with Control-IQ plus CGM: Following SAP, subjects will be utilizing the Tandem t:slim X2 with Control-IQ along with a Dexcom G6 continuous glucose monitor to control their blood glucose for 4 weeks. Subjects will be evaluated by actigraphy watch and by Ecological Momentary Assessments in approximately the final 14 days of the 4 week period.
Arm/Group | Older Adults:Sensor Augmented Pump (SAP) | Older Adults: Closed-Loop Control (CLC) | Young Children: SAP | Young Children: CLC
Number analyzed (Participants) | 15 | 15 | 13 | 13
percentage of time | 69.6 (14.2) | 79.6 (7.8) | 50.9 (12) | 69.2 (9.2)
Statistical Analysis 1: Comparison: Older Adults:Sensor Augmented Pump (SAP) vs Older Adults: Closed-Loop Control (CLC); Test type: Superiority; p = 0.002, t-test, 2 sided
Statistical Analysis 2: Comparison: Young Children: SAP vs Young Children: CLC; Test type: Superiority; p < 0.001, t-test, 2 sided

2. Secondary Outcome: Ecological Momentary Assessments
Description: Positive Moods were assessed using Ecological Momentary Assessments. Participants were asked a question on positive moods and answered on a Likert scale from 0 to 4 with a higher score indicating more positive mood. Scores were averaged from all evaluable completed assessment that were completed in the final 14 days of each study period.
Time Frame: Assessments will be administered during the final 14 days of each study period (sensor-augmented pump and closed-loop control).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Older Adults:Sensor Augmented Pump (SAP) | Older Adults: Closed-Loop Control (CLC) | Young Children: SAP | Young Children: CLC
Number analyzed (Participants) | 15 | 15 | 13 | 13
score on a scale | 2.42 (1.12) | 2.21 (0.93) | 2.45 (1.19) | 2.3 (1.37)

3. Secondary Outcome: Sleep Patterns
Description: Pittsburgh Sleep Quality Index (PSQI): a 10-item questionnaire assessment of sleep quality disturbances over the last month. Individual Items are rated on a 4 point Likert scale ranging from 0 to 3, which are then used to calculate a Global Score which can range from 0 to 21 with higher scores reflecting worse sleep quality. Parents completed the questionnaire for the young children cohort.
Time Frame: Assessments will be made at baseline and at the end of each study SAP (4 weeks) and CLC (4 weeks).
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Older Adults: Baseline; Young Children: Baseline: Baseline: prior to starting SAP
Arm/Group | Older Adults: Baseline | Older Adults:Sensor Augmented Pump (SAP) | Older Adults: Closed-Loop Control (CLC) | Young Children: Baseline | Young Children: SAP | Young Children: CLC
Number analyzed (Participants) | 15 | 15 | 15 | 13 | 13 | 13
score on a scale | 5.86 (3.01) | 5.71 (4.23) | 5.50 (3.11) | 4.38 (3.18) | 3.54 (2.6) | 3.62 (1.71)

ADVERSE EVENTS:
Time Frame: Duration of trial: approximately 10 weeks
Description: Adverse Event Collection was obtained for Older Adults and Children who were on the investigational CLC device. It was not obtained for parents who were not on the investigational CLC device.
Groups:
- Older Adults:SAP; Younger Children: SAP: SAP: Subjects will be utilizing their own insulin pumps (without automated insulin delivery) plus Dexcom G6 CGM to control their blood glucose for 4 weeks. Subjects will be evaluated by actigraphy watch and by Ecological Momentary Assessments in approximately the final 14 days of the 4 week period.
  e 4 week period.
  SAP: Subjects will wear their own personal insulin pump and will wear the study CGM (Dexcom G6).
- Older Adults: CLC; Younger Children: CLC: CLC with Control-IQ plus CGM: Following SAP, subjects will be utilizing the Tandem t:slim X2 with Control-IQ along with a Dexcom G6 continuous glucose monitor to control their blood glucose for 4 weeks. Subjects will be evaluated by actigraphy watch and by Ecological Momentary Assessments in approximately the final 14 days of the 4 week period.
  CLC: The Tandem t:slim X2 is an insulin pump with software (Control-IQ Technology) that helps regulate blood glucose more optimally, based on data received from the Dexcom G6 CGM.
Arm/Group | Older Adults:SAP | Older Adults: CLC | Younger Children: SAP | Younger Children: CLC
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15 | 0/13 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15 | 0/13 | 0/13
Other Adverse Events (participants affected / at risk) | 0/15 | 0/15 | 0/13 | 0/13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-01-23): https://cdn.clinicaltrials.gov/large-docs/81/NCT03674281/Prot_SAP_000.pdf
  • Informed Consent Form (2019-03-05): https://cdn.clinicaltrials.gov/large-docs/81/NCT03674281/ICF_001.pdf